CLINICAL TRIAL: NCT07296926
Title: Comparison of Efficacy of Distolingual Infiltration in Conjugation With Conventional Inferior Alveolar Nerve Block to Conventional Inferior Alveolar Nerve Block Alone for Extraction of Mandibular Third Molar
Brief Title: Distolingual Infiltration Verses Conventional Nerve Block in Mandibular Third Molar Extraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Watim Medical & Dental College (Other)
Responsible Party: Principal Investigator, aimen zafar, prinicpal investigator, Watim Medical & Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSG-2023-335-4631-A
Record Dates: First submitted 2025-11-26; First posted 2025-12-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pain (Visceral, Somatic, or Neuropathic)
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional nerve block injection (Active Comparator): Inferior alveolar and buccal nerve block using 2% lignocaine with adrenaline (1:80,000) without distolingual infiltration.
  Interventions: Procedure: Conventional Inferior Alveolar and Buccal Nerve Block
- conventional inferior alveolar with distolingual infilterate injection (Experimental): Inferior alveolar supplemented with distolingual infiltration using 2% lignocaine with adrenaline (1:80,000).
  Interventions: Procedure: Distolingual Infiltration plus Conventional Nerve Block

INTERVENTIONS:
Procedure: Conventional Inferior Alveolar and Buccal Nerve Block — Standard inferior alveolar and long buccal nerve block for mandibular third molar extraction.
  Arms: conventional nerve block injection
Procedure: Distolingual Infiltration plus Conventional Nerve Block — Distolingual infiltration (0.2 ml) administered in addition to conventional inferior alveolar during mandibular third molar extraction.
  Arms: conventional inferior alveolar with distolingual infilterate injection

SUMMARY:
This randomized controlled trial will compare the effectiveness of adding distolingual infiltration to conventional inferior alveolar and buccal nerve blocks for mandibular third molar extraction. A total of 120 patients will be allocated into two groups. Pain during flap elevation and bone guttering will be assessed using the Visual Analogue Scale.

DETAILED DESCRIPTION:
Mandibular third molar extraction is a common oral and maxillofacial surgery procedure that requires profound local anesthesia. Despite conventional inferior alveolar, lingual and buccal nerve blocks, the distolingual gingiva may remain non-anesthetized due to accessory innervation via the mylohyoid and other nerves. Distolingual infiltration may improve anesthesia in this area.

This randomized controlled trial will enroll 120 patients requiring mandibular third molar extraction. Participants will be randomized into two groups: conventional inferior alveolar and buccal nerve block (Group A) and the same technique with additional distolingual infiltration (Group B). Pain during mucoperiosteal flap elevation and bone guttering will be recorded on a 0-10 Visual Analogue Scale. The primary objective is to determine whether distolingual infiltration improves pain control compared to the conventional technique.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

  * Male and female
  * Age 18-45 years
  * Mandibular third molar impaction - all positions
  * Mandibular third molar impaction - all classes

Exclusion Criteria:

* ASA status III and above

  * Patients requiring multiple extractions in the same appointment
  * Allergy to lignocaine
  * Patients in whom adrenaline is contraindicated
  * Medically compromised individuals e.g. poorly controlled diabetes, hypertension

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Pain during mucoperiosteal flap elevation | During mucoperiosteal flap elevation on the day of surgery
  Pain intensity experienced during flap elevation will be assessed using the Visual Analogue Scale (VAS). This is a 0-10 point numerical scale where participants indicate the pain level experienced at the time of flap elevation.
  Measurement Tool:
  Visual Analogue Scale (VAS)
  Scale:
  * Minimum score: 0 (no pain)
  * Maximum score: 10 (worst possible pain)
  * Directionality: Higher scores indicate worse pain
Pain During Bone Guttering | During bone guttering on the day of surgery.
  Pain intensity during bone guttering will be recorded using the Visual Analogue Scale (VAS).
  Measurement Tool:
  Visual Analogue Scale (VAS)
  Scale:
  * Minimum: 0 (no pain)
  * Maximum: 10 (worst pain)
  * Higher scores = worse pain

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Aimen Zafar, Islamabad, Pakistan